CLINICAL TRIAL: NCT03805906
Title: Ultrasound-guided L5 Dorsal Ramus Block: Description and Validation of a Novel Technique
Brief Title: Ultrasound-guided L5 Dorsal Ramus Block
Acronym: USGL5DR
Status: Completed | Type: Observational
Sponsor: Montreal General Hospital (Other)
Collaborators: University of British Columbia (Other); Kelowna General Hospital (Other Government)
Responsible Party: Principal Investigator, Roderick Finlayson, Professor, Montreal General Hospital
Other Study IDs: 2018-19-061-H
Record Dates: First submitted 2019-01-13; First posted 2019-01-16 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Pain, Back
MeSH Terms: conditions — Back Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Primary group: Ultrasound-Guided L5 Dorsal ramus block
  Interventions: Procedure: L5 Dorsal ramus block

INTERVENTIONS:
Procedure: L5 Dorsal ramus block — Ultrasound-guided L5 dorsal ramus block

SUMMARY:
This study will examine the accuracy of an ultrasound-guided L5 dorsal ramus block technique.

DETAILED DESCRIPTION:
The lumbar facet joints have been implicated as a causal factor in 15 to 40% of patients suffering from chronic low back pain. Because physical examination and medical imaging have limited value in determining the source of pain, diagnostic blocks play an important role in the management of this common condition. Blocks of the L5 dorsal ramus (DR) are used to diagnosed pain originating from the L5-S1 facet joint, which is one of the most commonly implicated levels in patients with low back pain. Fluoroscopic guidance, which uses x-rays, is currently the standard imaging modality used to perform this block. Recently, ultrasound guidance has seen increasing use because of its greater accessibility and lack of ionizing radiation. Although USG has been shown to provide a high level of accuracy at other levels, the greater anatomical complexity found at the L5-S1 has hindered the development of a satisfactory L5 DR block technique. In this study the investigators will use fluoroscopic control to examine the accuracy of a novel ultrasound-guided approach to this block.

ELIGIBILITY:
Inclusion Criteria:

-Any consenting patient over 18 years of age with axial low back pain who requires a diagnostic L5 dorsal ramus block.

Exclusion Criteria:

* Inability to consent
* Iodine or lidocaine allergy,
* Pregnancy,
* Coagulopathy (as defined by an INR over 1.4, platelets under 100,000, or a documented bleeding disorder)
* Inability to visualize lumbosacral anatomy during an ultrasound pre- scan

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients suffering from chronic low back pain thought to involve the L5 dorsal ramus
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-01-12 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Block accuracy | Immediately post-injection
  contrast distribution

SECONDARY OUTCOMES:
Performance time | Perioperative
  Performance time as defined by the time the first image is acquired until the time the contrast injection is completed.
Number of needle passes | Procedure
  Number of needle passes required to perform block

CONTACTS AND LOCATIONS:
Locations (1):
- Kelowna General Hospital, Kelowna, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Etheridge JB, De Villiers F, Venter J, Squire P, Farnquist B, Finlayson RJ. Ultrasound-guided L5 dorsal ramus block: validation of a novel technique. Reg Anesth Pain Med. 2020 Mar;45(3):176-179. doi: 10.1136/rapm-2019-100783. Epub 2019 Oct 25. PMID 31653796